CLINICAL TRIAL: NCT03319810
Title: Proof of Concept of the Effect of Intravenous Immunoglobulin on Cerebral and Retinal Amyloid in Mild Cognitive Impairment Due to Alzheimer Disease
Brief Title: Effect of IVIG on Cerebral and Retinal Amyloid in Mild Cognitive Impairment Due to Alzheimer Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sutter Health (Other)
Responsible Party: Principal Investigator, Shawn Kile, M.D., Principal Investigator, Sutter Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIMR_Kile_IVIG POC
Record Dates: First submitted 2017-10-11; First posted 2017-10-24 (Actual); Results first posted 2019-04-16 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Mild Cognitive Impairment
Keywords: MCI, Alzheimer Disease, AD
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This is a single center, open label, proof of concept, out-patient study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- infusion of IVIG (Experimental)
  Interventions: Biological: Octagam 10%

INTERVENTIONS:
Biological: Octagam 10% — FDA approved human normal immunoglobulin solution ready for intravenous administration

SUMMARY:
This is a proof of concept study to determine if changes in brain amyloid levels are evident three months after infusion of 0.4 g/kg of IVIG every 14 days x 5 infusions. Amyloid levels will be measured by Florbetapir PET and retinal scan.

DETAILED DESCRIPTION:
Study design:

This is a single center, open label, proof of concept, out-patient study. Subjects will undergo Florbetapir PET and have retinal amyloid levels measured, receive an infusion of IVIG at 0.4 g/kg every 14 days for a total of five infusions, and repeat PET and retinal amyloid measures three months after the first infusion.

Subject population:

The study population will consist of male and female subjects diagnosed with mild cognitive impairment (MCI) due to Alzheimer disease (AD).

Estimated study duration:

The duration of each study subject is approximately 4 months, including one screening visit over a period of approximately 28 days, 5 days of infusions over a 2-month period of time, and a follow-up visit at 3 months after the first infusion.

Description of study drug:

Octagam is an FDA approved 10% human normal immunoglobulin solution ready for intravenous administration.

Study drug dosage:

The dose level of IVIG at 0.4 g/kg will be administered by IV infusion once every 14 days for two months.

Concomitant therapy:

Concomitant medications will be assessed at all study visits. Concomitant medications are prescribed or over-the-counter medications and should be consistent with the inclusion/exclusion criteria. Concomitant medication appropriate to the subject's condition may be prescribed during the course of the study with the exception of those listed above.

Routine vaccinations (i.e., flu vaccination) with commercially available therapeutics are permitted but must not be given within four weeks before or after the administration of the study drug.

Evaluations by visit:

Screening procedures at visit 1 will take place up to 28 days prior to Visit 2 (Day 1) dosing. Screening labs and assessments will be performed during the screening period. The first dose of study drug is administered on Day 1. Visits 2 through 6 have a ±1 day window and occur every 14 days over two months. The investigator will determine if a subject is suitable to continue following a missed infusion. Visit 7 has a ±7 day window.

All study screening data from Visit 1 including laboratory results must be reviewed for study eligibility prior to receiving first dose of study drug. Prior to infusion, a review of concomitant medications and AEs takes place. If the subject continues to be eligible for enrollment, the subject will be infused with study medication and will remain in the infusion clinic for at least 1 hour following the infusion for safety assessments on Visit 2 (Day 1), and 15 minutes for the subsequent visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 to <85 years.
2. Evidence of amyloid pathology on Florbetapir PET at screening.
3. Diagnosis of MCI due to AD based on NIA-AA criteria. (APPENDIX A)
4. MRI brain (with past 24 months) which shows evidence of mild hippocampal atrophy and/or bilateral parietal atrophy.
5. CDR score of 0.5
6. Mini-Mental State Examination (MMSE) score of 24-30, inclusive.
7. Rosen Modified Hachinski Ischemic score ≤4.
8. Receiving stable doses of medication(s) for the treatment of non-excluded medical condition(s) for at least 30 days prior to screening. Cholinesterase inhibitors and memantine are allowed if doses have stable been least 30 days prior to screening.
9. Agree to refrain from participating in any treatment or clinical trial targeting amyloid for the duration of the study.
10. Agree to refrain from taking any herbal supplement considered to enhance cognition unless approved by the investigator for the duration of the study.
11. Ability to attend all clinical visits and have an informant capable of accompanying the subject on specific clinic visits.
12. The subject's collaborative informant (support person) must be someone who has known the subject for at least 4 years and has had approximately 2 or more separate communications with the study participant per month (at least one of these communications in person).
13. Fluency in English and evidence of adequate premorbid intellectual functioning.
14. Adequate manual dexterity, visual, and auditory abilities to perform all aspects of the cognitive and functional assessments.
15. Venous access suitable for repeated infusions and phlebotomy.
16. In the opinion of the investigator, the subject and informant will be compliant and have a high probability of completing the study, including all scheduled evaluations and required tests.

Exclusion Criteria:

1. Has significant neurological disease other than MCI that in the opinion of the investigator may affect cognition.
2. History of clinically evident stroke or history of clinically significant carotid or vertebrobasilar stenosis or plaque.
3. History of seizures, excluding febrile seizures in childhood.
4. History of screening visit brain MRI scan indicative of any other significant abnormality, including but not limited to multiple microhemorrhages (2 or more), history or evidence of a single prior hemorrhage > 1 cm3, multiple lacunar infarcts (2 or more) or evidence of a single prior infarct > 1 cm3, evidence of a cerebral contusion, encephalomalacia, aneurysms, vascular malformations, subdural hematoma, or space occupying lesions of significance as determined by the PI (e.g., arachnoid cysts or brain tumors such as meningioma).
5. Brain MRI shows moderate or severe cortical or hippocampal atrophy.
6. Sensitivity to Florbetapir.
7. Other present/planned ionized radiation that, in combination with planned exposure to PET ligands for this study, would result in cumulative exposure that would exceed recommended limits.
8. Ophthalmologic condition that would interfere with retinal amyloid imaging.
9. Current presence of a clinically significant major psychiatric disorder (e.g., Major Depressive Disorder) according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV-TR) or symptom (e.g., hallucinations) that in the opinion of the investigator could affect the subject's ability to complete the study.
10. Current clinically significant systemic illness that is likely to result in deterioration of the subject's condition or affect the subject's safety during the study including but not limited to renal failure or myocardial infarction.
11. History of cancer within the last 5 years, with the exception of nonmetastatic basal cell carcinoma, and squamous cell carcinoma of the skin.
12. Uncontrolled hypertension (diastolic BP> 100 mmHg or systolic BP> 160 mmHg, sitting).
13. History or evidence of any clinically significant autoimmune disease or disorder of the immune system (e.g., Crohn's Disease, Rheumatoid Arthritis)
14. Clinically significant infection within the last 30 days (e.g., chronic persistent or acute infection (eg, upper respiratory infection [URI], urinary tract infection [UTI]).
15. Female subjects of childbearing potential.
16. Other clinically significant abnormality on physical, neurological, laboratory, vital signs or ECG examination (e.g., atrial fibrillation) that could compromise the study or be detrimental to the subject.
17. Weight greater than 120 kg (264 lbs).
18. Excessive smoking defined as more than 20 cigarettes per day.
19. History of alcohol or drug dependence or abuse as defined by DSM-IV criteria within the last 2 years.
20. Severe liver or kidney disease verified by the PI review of ALT, AST and creatinine.
21. Known coagulopathy, thrombosis, or low platelet count.
22. Hemoglobin less than 11 g/dL.
23. Known deficiency to IgA.
24. Positive serology for Hepatitis B or C, or HIV.
25. History of anti-amyloid treatment, immunotherapy, or other experimental treatment for MCI or Alzheimer disease.
26. Concurrent use of anticholinergic drugs including diphenhydramine.
27. Current use of anticoagulant medications (except the use of aspirin 325 mg/day or less, plavix, aggrenox, and persantine but not for stroke).
28. Concurrent use of opioid pain relievers and related synthetic derivatives.

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Kile, MD, Principal Investigator — Sutter Health; Carol Parise, PhD, Study Director — Sutter Health
Locations (1):
- Sutter Neuroscience Medical Group, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kile S, Au W, Parise C, Rose K, Donnel T, Hankins A, Chan M, Ghassemi A. IVIG treatment of mild cognitive impairment due to Alzheimer's disease: a randomised double-blinded exploratory study of the effect on brain atrophy, cognition and conversion to dementia. J Neurol Neurosurg Psychiatry. 2017 Feb;88(2):106-112. doi: 10.1136/jnnp-2015-311486. Epub 2015 Sep 29. PMID 26420886

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infusion of IVIG
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infusion of IVIG
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.30 (5.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Standard Uptake Value Ratio (SUVr) [Mean (Standard Deviation); unit: standard uptake value ratio] — SUVr is the ratio of activity per unit volume of a region of interest to the activity per unit whole body volume.
  standard uptake value ratio | 1.57 (0.16)

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline Standard Uptake Ratio Values (SUVr) of Florbetapir PET at 3 Months
Description: Amyloid deposition in the brain is thought to lead to the development of cognitive decline and conversion to AD. Each participant's amyloid burden can also be quantified through the computation of a Standard Uptake Value ratio (SUVr).
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: standard uptake value ratio
Arm/Group | Infusion of IVIG
Number analyzed (Participants) | 5
standard uptake value ratio | -3.83 (2.84)

2. Primary Outcome: Change in Baseline Retinal Amyloid Imaging (RAI) at 3 Months
Description: This is a noninvasive imaging technique that can detect amyloid-beta deposition in the retinas of the eye.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: autofluorescent spot count
Arm/Group | Infusion of IVIG
Number analyzed (Participants) | 5
autofluorescent spot count
  Right Eye | -33.00 (68.52)
  Left Eye | -55.75 (46.95)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Infusion of IVIG
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infusion of IVIG (N=5)
dizziness (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT03319810/Prot_SAP_000.pdf